CLINICAL TRIAL: NCT03648697
Title: A Pilot Study of EBV-TCR-T(YT-E001) in NPC Patients
Brief Title: EBV-TCR-T（YT-E001）for Patients With EBV-positive Recurrent or Metastatic NPC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fujian Cancer Hospital (Other Government)
Collaborators: China Immunotech (Beijing) Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HXYT-001
Record Dates: First submitted 2018-08-24; First posted 2018-08-27 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Cell Count; fludarabine; Cyclophosphamide

STUDY DESIGN:
Intervention Model Description: Single arm, open label, single dose phase I/II study of safety and efficacy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EBV-TCR-T cells(YT-E001) (Experimental): EBV-TCR-T (YT-E001) cells are prepared via lentiviral infection. 6-10 days prior to infusion of TCR-T cells (YT-E001), subjects receive fludarabine at dose 30mg/m2/day for 4 days and cyclophosphamide treatment at dose 30mg/kg/day for 2 days and take a rest for one day before infusion.
  A single dose of EBV-TCR(YT-E001) transduced T cells (about 2×108) will be intravenously (i.v.) administered.
  Interventions: Biological: EBV-TCR-T (YT-E001) cells

INTERVENTIONS:
Biological: EBV-TCR-T (YT-E001) cells — EBV-TCR-T (YT-E001) cells are prepared via lentiviral infection. 6-10 days prior to infusion of TCR-T cells (YT-E001), subjects receive fludarabine at dose 30mg/m2/day for 4 days and cyclophosphamide treatment at dose 30mg/kg/day for 2 days and take a rest for one day before infusion.
  Patients, who receive an infusion of YT-E001, will remain in the hospital to be monitored for adverse events until they have recovered from the treatment. Patients will have frequent follow-up visit to monitor the persistence of modified T cells and efficacy of the treatment.
  Other Names: Fludarabine; Cyclophosphamide

SUMMARY:
TCR-T cell therapy experienced a breakthrough for treating tumors in recent years. Phase I / II trial of NY-ESO-1-specific TCR-T treatment for synovial sarcoma and melanoma conducted by the Rosenberg team at the National Cancer Institute showed that 61% Synovial cell sarcoma and 55% melanoma had therapeutic responses. These and lots of clinical achievements indicate that TCR-T cell therapy can target a variety of tumors including solid tumors without any severe side effects found in CAR-T trials.

Nasopharyngeal carcinoma (NPC), a kinds of head-neck malignant tumor, which used to appear mostly in southern China (especially in Fujian and Guangdong and Guangxi provinces). Most patients with NPC show evidence of infection with the Epstein Barr virus (EBV) before or at the time of their diagnosis. EBV is found in the cancer cells of almost all patients with advanced stage NPC, and play a role in causing and inducing the disease program and development. The cancer cells infected by EBV are able to hide from the body's immune system and escape destruction. We want to see if EBV antigen special T cells (YT-E001) could recognize and kill special parts of EBV infected cells, and finally inhibit the tumor recurrence or metastasis of NPC patients.

This study will focus on the NPC highly expressed EBV antigen such as LMP1, LMP2 and EBNA1，the high affinity TCR target the above EBV antigen were screened from the healthy donor using the sorting and single cell cloning technique. Then, using the lentivirus to transduce the TCR gene to the autologous T cells.

This study will investigate the safety and tolerability of EBV-TCR-T cell therapy in subjects with NPC who had received prior therapy for their disease but their disease has progressed or relapsed.

The chemotherapy we will use for lymphodepletion is a combination of cyclophosphamide and fludarabine. Cyclophosphamide and fludarabine are the chemotherapy agents most commonly used for lymphodepletion in immunotherapy clinical trials.

DETAILED DESCRIPTION:
This Phase I/II study is designed as single dose pilot trial evaluating the safety and of EBV-TCR-TT cell therapy in subjects with NPC who have received prior therapy for their disease but the disease has progressed or relapsed. Anti-tumor activity and other exploratory objectives will be assessed. Subjects enter from a Screening Protocol and are positive for HLA- A02:01/24:02/11:01, and EBV serum positive. Subjects will receive cytoreductive chemotherapy with cyclophosphamide and fludarabine on days -6 and -4 followed by infusion of dose of about 2×108 EBV-TCR-T(YT-E001).

Subjects will stay in hospital for safety and efficacy assessment daily from T cell infusion (Day 0) through Day 7, and then weekly until week 4 and then at 8 weeks every 8 weeks until progression of their disease or the end or termination of trial.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old;
2. Sign an informed consent before undertaking any trial-related activities;
3. NPC patients diagnosed by licensed pathologist, EBV DNA copy number >500.
4. Received at least one run of standard therapy (surgery, chemo, radiation and targeted therapy) or first line and second line treatment failure;
5. HLA-A*0201/2402/1101;
6. ECOG score 0-2；Life expectancy is longer than 3 months;
7. No Chinese herbal medicine usage within 4 weeks before enrollment;
8. Lab test results meet the following requirements:

   White blood cell count≥4.0×109/L; ANC≥1.5 ×109/L; PLT≥100 ×109/L; Hemoglobin≥90g/L; Prothrombin time or INR ≤1.5× normal upper limit, except taking anticoagulant therapy; PTT≤1.5× normal upper limit；AST≤3×ULN; ALT≤3×ULN; ALP≤3×ULN; TBIL≤1.5×ULN。
9. Levels of calcium, potassium, and magnesium in serum are within the normal range;
10. Pregnancy test is negative for female subjects with reproductive capability before participating the study Female subjects must consent using birth control during the study or prohibit any homo or heterosexual behavior;
11. Can regularly visit the research institutions for tests, evaluations, and monitoring throughout the study period.

Exclusion Criteria:

1. Received major surgery, conventional chemotherapy, large-area radiotherapy, immune therapy or any biological anti-tumor therapy within 4 weeks prior to the study;
2. Allergic to any components of the therapy;
3. Never recovered to <2 grade CTCAE from prior surgery or treatment-related adverse events;
4. With two or other types of primary solid tumors;
5. Poorly managed hypertension (systolic blood pressure >160 mmHg and / or diastolic blood pressure > 90 mmHg) or clinically significant(for example, active) cardiovascular and cerebrovascular diseases such as cerebrovascular incident (within 6 months prior to signing the informed consent), myocardial infarction (within 6 months prior to signing the informed consent), unstable angina, grade II or above heart failure, Congestive, or severe arrhythmia can not be controlled by medication or has a potential impact on the study;
6. With other serious organic disease and/or mental illness;
7. With systemic active infections that need treatments, including active tuberculosis, HIV/HBV/HCV- positive or clinically active hepatitis A, B and C;
8. With autoimmune diseases: such as a history of inflammatory bowel disease (IBD) or other autoimmune diseases determined by the investigator to be unsuitable for the study (e.g. systemic lupus erythematosus (SLE), vasculitis, invasive pulmonary disease);
9. Within 4 weeks prior the infusion, received chronic systemic steroid cortisone, Hydroxyurea, immunomodulatory treatment (for example: Interleukin 2, alpha or gamma interferon, GCSF, cyclosporine etc.);
10. History of organ allografts, autologous / allogeneic stem cell transplantation, and renal replacement therapy;
11. With central nervous system metastasis.
12. With uncontrolled diabetes, pulmonary fibrosis, interstitial lung disease, acute lung disease, or liver failure;
13. Pregnant or lactating female patients;
14. Received concomitant medication prohibited by the protocol;
15. With any medical condition or disease determined by the investigators that may be detrimental to this trial;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-10-10 (Actual); Primary Completion 2021-10-08 (Estimated); Study Completion 2021-10-10 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events | 60 days
  To evaluate the safety and feasibility of the administration of EBV-TCR transduced T cells(YT-E001) in patients with EBV+ NPC.

SECONDARY OUTCOMES:
Number of participants with clinical responses | 1 YEAR
  To evaluate the efficacy of EBV positive NPC patients treated with EBV antigen specific affinity-enhanced TCR transduced autologous T cell therapy(YT-E001).

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Cancer Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No